CLINICAL TRIAL: NCT02472106
Title: Impact of Postdilatation With the InterValve V8 Aortic Valvuloplasty Balloon Following Medtronic CoreValve or Other Self-Expanding TAVI Procedure (PostCorE)
Brief Title: Impact of Postdilatation With the InterValve V8 Aortic Valvuloplasty Balloon Following TAVI Procedure
Acronym: PostCorE
Status: Completed | Type: Observational
Sponsor: InterValve, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1302-001
Record Dates: First submitted 2015-05-28; First posted 2015-06-15 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve; TAVI; Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Post-dilatation — Post-dilatation in self-expanding TAVI device procedures

SUMMARY:
This study is designed to monitor the safety and performance of the V8 balloon when used as a postdilatation balloon in self-expanding Transcatheter Aortic Valve Implantation (TAVI) device procedures. The study product is CE marked for balloon aortic valvuloplasty (BAV), and is being investigated for an expanded intended use.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, single arm open-label clinical study involving up to 5 centers and a minimum of 20 subjects. Up to 50 subjects may be enrolled in this study. The first 3 post-dilatation procedures for each investigator will be considered roll-ins and not included in the main study analyses. Subjects will exit the study at hospital discharge or 7 days post treatment, whichever comes first. The expected duration of the clinical investigation is approximately 6 months.

Subjects implanted with the CoreValve or other commercially available self-expanding TAVI and with the use of the V8 as a postdilatation balloon may be enrolled in this study. The subject will exit the study after the predischarge ECHO where the Paravalvular Leak (PVL) measurements are taken or resolution of a V8 related AE (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe symptomatic aortic stenosis (AS) indicated and scheduled for a transcatheter aortic valve implant (TAVI) with the Medtronic CoreValve or another self-expanding TAVI device.
* The TAVI device size is determined preoperatively with CTA according to standard guidelines. Patients may undergo transfemoral, subclavian, or transaortic approach.
* Balloon postdilatation (BPD) is carried out after CoreValve or other self-expanding TAVI device implantation if, based on operator's judgment, BPD is indicated because of presence of paravalvular leak (PVL).
* Hemodynamically stable for 3 - 10 minutes after the TAVI procedure.
* Probable survival to hospital discharge.
* Subject is competent, willing to comply with evaluations, understands risks, benefits and alternatives and has signed the Informed Consent Form.

Exclusion Criteria:

* Cardiogenic shock, as defined by a consistent systolic blood pressure <80 mmHg off vasopressors or <90 mmHg on vasopressors.
* PVL occurring secondary to excessively high or low valve positioning.
* Trauma or significant structural damage to underlying native tissue calls for emergent intervention or threatens long-term outcome prior to the BPD.
* Patients receiving two valves (i.e. aortic THV valve in valve).
* Patients with AS secondary to congenital valve disease including bicuspid aortic valve.
* PVL occurring due to TAVI device under sizing. Example of determining the undersizing is to calculate the Cover Index which represents the percent of over sizing of the nominal transcatheter heart valve (THV) area compared to the measured native valve annulus area. Under sizing is defined as TAVI screening CTA with a pre procedure cover index by area of <5%.
* Vulnerable subjects and any subjects incapable of giving consent, including patients with incurable diseases, patients in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, minors, and subjects with cognitive impairment, such as persons with a mental illness or dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic - Patients at each enrolling clinic who are to be treated with the Medtronic CoreValve or other self-expanding TAVI device are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Efficacy Endpoint: V8 Device Performance | Intra-Procedure
  Rate of successful V8 balloon fixation within the TAVI prosthesis: during rapid ventricular pacing, proximal and distal balloon segments are securely fixed on either side of the native aortic valve annulus following inflation
Safety Endpoint: Serious Adverse Events (SAE) | Intra-procedure until discharge or 7 days post-procedure, whichever comes first. (Typical discharge is expected to be within 7 days.)
  The composite of SAEs as defined by the Valve Academic Research Consortium (VARC II)

SECONDARY OUTCOMES:
Efficacy Endpoint: Degree of Paravalvular Leak (PVL) | Intra-Procedure
  PVL determined by collating as many data points as possible using TTE, TEE, aortic root angiography, and/or hemodynamic measurements
Efficacy Endpoint: Procedural Parameter - V8 Dimension | Intra-Procedure
  Size of V8(s) used during procedure
Efficacy Endpoint: Procedural Parameter - CoreValve Dimension | Intra-Procedure
  Size of CoreValve(s) used during procedure
Efficacy Endpoint: Procedural Parameter - Aortic Valve Measurement | Intra-Procedure
  Aortic Valve measurements performed during procedure
Safety Endpoint: 24hr Complication | 24 hours post-procedure
  AE(s) defined in protocol attributable to V8 balloon post-dilatation (BPD) procedure